CLINICAL TRIAL: NCT05680168
Title: Efficacy of Extracorporeal Magnetic Stimulation, Pelvic Floor Muscle Exercise, and Combination of Both in Management of Post Radical Prostatectomy Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Efficacy of Extracorporeal Magnetic Stimulation, Pelvic Floor Muscle Exercise, and Combination of Both in Management of Post Radical Prostatectomy Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad General Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmed Albakr, Principal Investigator, Hamad General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC0122185
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Post Radical Prostatectomy Urinary Incontinence
Keywords: Radical prostatectomy; Magnetic stimulation; pelvic floor exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Extracorporeal Magnetic stimulation (Active Comparator): Group (A): will receive rehabilitation program with exposure to ExMS, Patients will receive regular sessions of electromagnetic stimulation using Magneto STYM device, (Iskra medical d.o.o, Slovenia). Each session will last for 20 minutes. Patients will receive three weekly sessions for total of 20 sessions starting one month after catheter removal.
  Interventions: Device: Extracorporeal electromagnetic stimulation
- Group B: Extracorporeal Magnetic stimulation and pelvic floor exercises (Active Comparator): Group (B): This group will receive a rehabilitation program depending ExMS with the protocol described above. In addition, this group will be advised for pelvic floor muscle training in serial training sessions with our therapist for PME.
  Interventions: Device: Extracorporeal electromagnetic stimulation; Behavioral: Pelvic floor exercises
- Group C: Pelvic floor exercises (Active Comparator): Group (C): This will be the control group. This group will be advised to do PME only. The pelvic floor exercises will consist of advice to the patients to contract the anal sphincter muscles in successive way as if holding flatus. The pelvic floor muscle training schedule and therapist in group B and group C will be the same.
  Interventions: Behavioral: Pelvic floor exercises

INTERVENTIONS:
Device: Extracorporeal electromagnetic stimulation — Electromagnetic stimulation using Magneto STYM device, (Iskra medical d.o.o, Slovenia).
  Arms: Group A: Extracorporeal Magnetic stimulation; Group B: Extracorporeal Magnetic stimulation and pelvic floor exercises
Behavioral: Pelvic floor exercises — Pelvic floor muscle training in serial training sessions with our therapist
  Arms: Group B: Extracorporeal Magnetic stimulation and pelvic floor exercises; Group C: Pelvic floor exercises

SUMMARY:
Urinary incontinence is one of the most common complications of radical prostatectomy. Multiple prevention and treatment modalities have been proposed in the management of post prostatectomy urinary incontinence. This is a randomized controlled comparative study to evaluate the efficacy of extracorporeal magnetic stimulation alone and combined with pelvic floor muscle exercise versus pelvic floor muscle exercise alone in the management of post radical prostatectomy urinary incontinence. This study is expected to be performed over 7 years. The study population will be all male patients who are prepared for radical prostatectomy under urology department in HMC and were referred to voiding dysfunction for preoperative counselling and postoperative rehabilitation. Patients will be randomized into one of three treatment groups. The first group will receive sessions of extracorporeal magnetic field stimulation only. The second group will receive extracorporeal magnetic stimulation in addition to pelvic floor muscle exercise. The third group will receive pelvic floor muscle exercise only. The recruitment phase will take 3 years. Patients will be followed for 18 months for the course of urinary incontinence symptoms, severity of urinary incontinence on 1-hour pad test, urodynamic leak point pressure and the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) and the ICIQ quality of life (QOL) score. This study is proposed to reveal strong evidence on the efficacy of extracorporeal magnetic stimulation on the management of post radical prostatectomy urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include all adult male patients 18 years of age and above, with localized prostate cancer of low or intermediate risk disease who chose definitive treatment with radical prostatectomy either through open radical retropubic prostatectomy (RRP) or through robotic assissted laparoscopic radical prostatectomy (RALP) as first line for treatment and had the surgery under Hamad General Hospital urology department care.

Exclusion Criteria:

* Patients with high risk , locally advanced or metastatic prostate cancer at time of diagnosis
* Patients with low to intermediate risk prostate cancer who received chemo or radiotherapy then had salvage surgery
* Patients with urinary incontinence or diagnosed overactive bladder before radical prostatectomy.
* Patients with complicated surgery resulting in anastomotic leak, prolonged catheterisation more than 3 weeks, reinsertion of catheter due to retention of urine.
* Patients who refuse to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
One hour pad test | 18 months from the start of intervention
  Measuring the weight of an incontinence pad used for one hour to detect the volume of urinary leakage in one hour assessed at 6 points of follow up
the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | 18 months from the start of intervention
  Questionnaire administered at 6 points of follow up
Urodynamic leak point pressure. | 1 day (Once) after 6 weeks of the start of rehabilitation process
  Urodynamic study to evaluate the bladder dynamics and its response to radical prostatectomy and its response to rehabilitation

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire quality of life score | 18 months from the start of intervention
  Questionnaire administered at 6 points of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Ambulatory Care Center, Doha, Qatar